CLINICAL TRIAL: NCT01185314
Title: A Molecular Epidemiology Study in Asian Patients With Advanced Non-small Cell Lung Cancer (NSCLC) of Adeno Histology to Assess Epidermal Growth Factor Receptor (EGFR) Mutation Status
Brief Title: To Study the Changes in Protein in Lung Cells of Asian Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: PIONEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Gerard Lynch, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D7913L00086
Record Dates: First submitted 2010-08-16; First posted 2010-08-19 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC, EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): EGFR mutation testing
  Interventions: Procedure: Testing for mutation status

INTERVENTIONS:
Procedure: Testing for mutation status — EGFR mutation test

SUMMARY:
The purpose of this study is to study the changes in protein in lung cells of Asian patients with advanced non small cell lung cancer.

DETAILED DESCRIPTION:
A molecular epidemiology study in Asian patients with advanced NSCLC of adeno histology to assess EGFR mutation status.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologically confirmed advanced Non small cell lung cancer of adeno histology NSCLC treatment naive Availability of cancer tissue or cytology sample

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study Previous enrollment in the present study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1270 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
EGFR mutation status of Asian patients with advanced NSCLC | Samples will be tested after informed consent. Mutation results will be available within 1-3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Yeoman, MBBS, MFPM, Study Director — AstraZeneca; Robin Meng, MD, PhD, Study Chair — AstraZeneca Taiwan; Yang Pan-Chyr, MD, PhD, Principal Investigator — National Taiwan University College of Medicine
Locations (36):
- China (12):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
- Research Site, Hong Kong, Hong Kong, Hong Kong
- India (7):
  - Research Site, Chennai, Chennai
  - Research Site, Vadodara, Gujarat
  - Research Site, Kochi, Kerala
  - Research Site, Kolkata, Kolkata
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Rohini, National Capital Territory of Delhi
- Philippines (5):
  - Research Site, Cebu City
  - Research Site, City of Taguig
  - Research Site, Manila
  - Research Site, Pasay
  - Research Site, Quezon City
- Taiwan (6):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok, Bangkok
  - Research Site, Songkhla, Changwat Songkhla
  - Research Site, Chiang Mai, Chiang Mai
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City